CLINICAL TRIAL: NCT06885827
Title: Interventional Vitamin Mix Glaucoma Study (IVMGS) - A Prospective, Randomized, Two-Arm, Single-Center Study Protocol in Existing Glaucoma Patients.
Brief Title: Vitamin Mix (B6, B9, B12, And Choline) For Glaucoma Patients
Acronym: IVMGS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Collaborators: St. Erik Eye Hospital (Other)
Responsible Party: Principal Investigator, Rune Brautaset, Professor, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2023-06239-01
Record Dates: First submitted 2025-03-10; First posted 2025-03-20 (Actual); Last update posted 2025-04-29 (Actual); Status verified 2025-04

CONDITIONS: Open-angle Glaucoma; Pseudoexfoliation Glaucoma
Keywords: methyl donor supplementation; glaucoma; neuroprotection; randomized clinical trial; open-label; B6; B9; choline; visual field; optical coherence tomography; electroretinogram
MeSH Terms: conditions — Glaucoma, Open-Angle; Exfoliation Syndrome; Glaucoma | interventions — Standard of Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention (Active Comparator): Participants in this arm receive both the Vitamin B-mix supplement and standard glaucoma care.
  Interventions: Dietary Supplement: Vitamin B-mix
- Controls (Active Comparator): Participants in this arm receive standard glaucoma care only.
  Interventions: Other: Standard Care

INTERVENTIONS:
Dietary Supplement: Vitamin B-mix — Daily oral supplementation with:
  Vitamin B6 (pyridoxine, 25 mg), 1 capsule Vitamin B9 (folic acid, 400 µg) + Vitamin B12 (cyanocobalamin, 1 mg), 2 capsules.
  Choline (choline bitartrate, 500 mg), 2 capsules Administered alongside standard glaucoma care.
  Arms: Intervention
Other: Standard Care — Usual glaucoma management (e.g., monitoring and/or IOP-lowering treatments) without additional supplementation.
  Arms: Controls

SUMMARY:
This study aims to determine whether a combination of vitamins (B6, B9, B12, and choline) can help protect the eyes of people with glaucoma and slow vision loss. The study will assess whether these vitamins support retinal cells and maintain or improve their function.

Adults aged 18 and older with primary open-angle glaucoma (including normal-tension glaucoma) or pseudoexfoliation glaucoma, and those with mild to moderate glaucoma, may be eligible. Participants must meet specific medical criteria and cannot take additional vitamin supplements during the study.

Participants will be randomly assigned to one of two groups: one group will take a daily vitamin supplement (B6, B9, B12, and choline) for one year, along with standard glaucoma care, while the other will continue standard care without extra vitamins. The vitamins used are well tolerated at selected doses, with possible mild side effects such as an upset stomach or tingling sensations. They will visit the clinic five times over 12 months (at the start, and at 3, 6, 9, and 12 months) for routine eye tests, including measuring eye pressure, checking vision and visual fields, taking scans of the eye's nerve layers (OCT), and completing an electroretinogram (ERG) to assess retinal function. Blood samples will also be collected.

If the vitamins are effective, this could provide an additional strategy alongside current eye pressure lowering treatments to reduce vision loss.

ELIGIBILITY:
Eligibility Criteria

Inclusion Criteria:

Patients with the following characteristics will be eligible for inclusion in the trial:

* 18 years or older at the time of inclusion
* Diagnosis of Primary Open-Angle Glaucoma (POAG), Normal Tension-Glaucoma (NTG) or Pseudoexfoliation Glaucoma (PEXG) in one or both eyes diagnosticed by an ophthalmologist.
* Best corrected Snellen VA of 0.3 or better in the study eye(s)
* Two or more reliable VF tests with less than 15% false positives

Exclusion Criteria:

Patients who meet any of the following criteria will be excluded from participation in the study:

* Visual field damage worse than -16dB in the study eye(s)
* Eye pressure greater than 35 mmHg in study eye(s) on either of two measurement occasions or a mean pressure of 30 mmHg over two occasions
* Any disease affecting retinal function
* Neurological or other non-glaucomatous conditions that may affect the visual field
* Inability to perform visual field examination
* Unwillingness to stop any intake of multivitamins or B vitamin substances
* Known allergy or intolerance to B-vitamins
* Previous eye surgery, except for uncomplicated cataract surgery
* Pregnant or breastfeeding women
* Women of childbearing potential who do not use reliable contraception
* Any disease or condition likely to prevent long-term follow-up
* Cancer diagnosis within the last 5 years (except treated squamous cell carcinoma)
* History of liver disease or stomach ulcers
* Inability to understand and speak Swedish or English

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-03-31 (Actual); Primary Completion 2027-03-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Change in photopic negative response (PhNR) on electroretinography (ERG) | Baseline, third month and twelfth month.
  The primary outcome is the change in retinal function as measured by the PhNR on ERG over a 12-month period.

SECONDARY OUTCOMES:
Changes to retinal structure | Baseline, third month and twelfth month.
  Measurement of retinal nerve fiber layer (RNFL) and ganglion cell layer-inner plexiform layer (GCL-IPL) thickness via OCT.
Change in Visual Field Index (VFI) | Baseline, third month, and twelfth month.
  Changes in Visual Field Index (VFI) assessed by automated perimetry. Unit of Measure: Percentage (%).
Blood biomarkers | Baseline, third month and twelfth month.
  Analysis of blood metabolomic profiles and global DNA methylation levels to evaluate systemic effects of the intervention.
Intraocular Pressure (IOP) | From baseline to twelfth months.
  Measured using ICare tonometer.
Change in Best Corrected Visual Acuity (BCVA) | From baseline to twelfth months.
  Measured using the Early Treatment Diabetic Retinopathy Study (ETDRS) letter score.
  Minimum Value: 0 (worst visual acuity). Maximum Value: 100 (best visual acuity) Interpretation: Higher scores indicate better visual acuity.
Change in Mean Deviation (MD) | Baseline, third month, and twelfth month.
  Changes in Mean Deviation (MD) assessed by automated perimetry. Unit of Measure: Decibels (dB).
Change in Pattern Standard Deviation (PSD) | Baseline, third month, and twelfth month.
  Changes in Pattern Standard Deviation (PSD) assessed by automated perimetry. Unit of Measure: Decibels (dB)

CONTACTS AND LOCATIONS:
Overall Officials: Rune Brautaset, Professor of Optometry, Principal Investigator — Karolinska Institutet
Locations (2):
- Sweden (2):
  - St Eriks Ögonsjukhus, Stockholm, Stockholm County
  - Karolinska institutet, The Division of Eye and vision., Stockholm, Stockholm County

IPD SHARING:
Plan to Share IPD: Undecided
We aim to share pseudonymized individual participant data that underlie results in a publication in accordance with institutional regulations.

REFERENCES:
- [Derived] Golpour N, Hui F, Nilsson M, Svensson J, Brautaset RL, Tribble JR, Williams PA. Interventional Vitamin Mix Glaucoma Study (IVMGS): study protocol for a prospective, randomized, two-arm, single-center trial in existing glaucoma patients. Trials. 2025 Oct 13;26(1):403. doi: 10.1186/s13063-025-09168-z. PMID 41084053